CLINICAL TRIAL: NCT01610284
Title: A Phase III Randomized, Double Blind Placebo Controlled Study of BKM120 With Fulvestrant, in Postmenopausal Women With Hormone Receptor-positive HER2-negative Locally Advanced or Metastatic Breast Cancer Which Progressed on or After Aromatase Inhibitor Treatment
Brief Title: Phase III Study of BKM120/Placebo With Fulvestrant in Postmenopausal Patients With Hormone Receptor Positive HER2-negative Locally Advanced or Metastatic Breast Cancer Refractory to Aromatase Inhibitor
Acronym: BELLE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBKM120F2302; 2011-005524-17 (EudraCT Number)
Record Dates: First submitted 2012-05-11; First posted 2012-06-04 (Estimated); Results first posted 2020-06-18 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Hormone receptor positive; HER2-negative; Metastatic; Locally advanced; PI3K; Fulvestrant; Refractory; Aromatase inhibitor
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Fulvestrant; NVP-BKM120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BKM120 100mg + Fulvestrant (Experimental): BKM120 100 mg per day and fulvestrant given until progression or as described in the protocol.
  Interventions: Drug: Fulvestrant; Drug: BKM120
- Placebo + Fulvestrant (Placebo Comparator): BKM120 matching placebo daily and fulvestrant given until progression or as described in the protocol.
  Interventions: Drug: Fulvestrant; Drug: BKM120 matching placebo

INTERVENTIONS:
Drug: Fulvestrant — Intramuscular fulvestrant 500 mg (Day 1 and Day 15 of Cycle 1 and Day 1 of every cycle thereafter)
Drug: BKM120 — BKM120 100 mg once daily
  Arms: BKM120 100mg + Fulvestrant
Drug: BKM120 matching placebo — BKM120 matching placebo, once daily
  Arms: Placebo + Fulvestrant

SUMMARY:
This study was a multi-center, randomized, double-blind, placebo controlled Phase III study to determine the efficacy and safety of treatment with buparlisib plus fulvestrant versus fulvestrant plus placebo in postmenopausal women with hormone Receptor-positive (HR-positive), human epidermal growth factor receptor 2-negative (HER2-negative), locally advanced or metastatic breast cancer (MBC) whose disease has progressed on or after aromatase inhibitor (AI) treatment.

DETAILED DESCRIPTION:
Patients were randomized (1:1) to receive buparlisib (100 mg/day) or placebo with fulvestrant (500 mg); randomization was stratified by PI3K pathway activation status (activated, non-activated, unknown determined in archival tumor tissue) and visceral disease status (present or absent). Tumor evaluation was performed 6 weeks after the randomization date and then every 8 weeks until radiological progression (based on Response Evaluation Criteria In Solid Tumors [RECIST] version 1.1).

Novartis made the decision not to pursue further development of buparlisib and to terminate the ongoing studies in the program. Accordingly, on 19-Dec-2016, Novartis notified all the Investigators about the decision not to pursue further development of buparlisib in Breast Cancer. As a result, the CBKM120F2302 study was terminated on 19-Apr-2019 (last subject last visit).

ELIGIBILITY:
Key Inclusion Criteria:

* Locally advanced or metastatic breast cancer
* HER2-negative and hormone receptor-positive status (common breast cancer classification tests)
* Postmenopausal woman
* A tumor sample must be shipped to a Novartis designated laboratory for identification of biomarkers (PI3K activation status)
* Progression or recurrence of breast cancer while on or after aromatase inhibitor treatment
* Measurable disease or non measurable disease bone lesions in the absence of measurable disease as per RECIST 1.1
* Adequate bone marrow and organ function defined by laboratory values

Key Exclusion Criteria:

* Previous treatment with PI3K inhibitors, AKT inhibitors, mTOR inhibitor or fulvestrant
* More than one prior chemotherapy line for metastatic disease
* Symptomatic brain metastases
* Increasing or chronic treatment (> 5 days) with corticosteroids or another immunosuppressive agent
* Active heart (cardiac) disease as defined in the protocol
* Certain scores on an anxiety and depression mood questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1147 (Actual)
Dates: Start 2012-08-07 (Actual); Primary Completion 2015-04-29 (Actual); Study Completion 2019-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (239):
- United States (61):
  - University of South Alabama / Mitchell Cancer Institute Deptof Mitchell Cancer Inst(2), Mobile, Alabama
  - Arizona Oncology Associates Dept of Oncology, Phoenix, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Shapiro and Stafford and Yee and Polanski Study Coordinator, Arcadia, California
  - Cancer Care Associates Dept.ofCancerCareAssoc., Fresno, California
  - St. Jude Heritage Medical Group Virginia Crosson Cancer Center, Fullerton, California
  - University of California San Diego - Moores Cancer Center UCSD 3, La Jolla, California
  - Los Angeles Hematology/Oncology Medical Group LA Cancer Network, Los Angeles, California
  - USC Kenneth Norris Comprehensive Cancer Center Dept.ofNorrisCompCancerCtr (3), Los Angeles, California
  - University of California at Los Angeles Dept. of UCLA, Los Angeles, California
  - Ventura County Hematology and Oncology PMK Medical Group, Oxnard, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Santa Barbara Hematolgy Oncology Medical Group, Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - St Joseph Heritage Healthcare Dept. of RRMG (4), Santa Rosa, California
  - Granada Hills Cancer Center, Valencia, California
  - Kaiser Permanente Northwest Kaiser, Denver, Colorado
  - Rocky Mountain Cancer Centers RMCC, Greenwood Village, Colorado
  - Memorial Regional Cancer Center MRCC, Hollywood, Florida
  - Cancer Specialists of North Florida SC - F2302, Jacksonville, Florida
  - University of Miami Univ Miami 2, Miami, Florida
  - MD Anderson Cancer Center - Orlando MD Orlando, Orlando, Florida
  - Georgia Cancer Specialists SC, Decatur, Georgia
  - North Shore University Health System, Evanston, Illinois
  - Cadence Health, Geneva, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland Niles, Multiple Locations, Illinois
  - Cancer Center of Kansas CCK, Wichita, Kansas
  - Mercy Medical Center Mercy Medical SC, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center Johns Hopkins Med Sidney/John Hopkins, Baltimore, Maryland
  - Frederick Memorial Hospital Fred. Mem. Hosp., Frederick, Maryland
  - Maryland Oncology Hematology, P.A. SC, Rockville, Maryland
  - Massachusetts General Hospital SC, Boston, Massachusetts
  - West Michigan Cancer Center Dept of Oncology, Kalamazoo, Michigan
  - Hematology and Oncology Association at Bridgepoint Hem Onc Bridgepoint, Tupelo, Mississippi
  - Washington University School of Medicine Regulatory, St Louis, Missouri
  - Hackensack Meridian Health, Brick, New Jersey
  - The Valley Hospital / Luckow Pavillion, Paramus, New Jersey
  - Clinical Research Alliance SC-2, Lake Success, New York
  - Memorial Sloan Kettering Dept Onc, New York, New York
  - University of Rochester Medical Center Univ Rochester, Rochester, New York
  - Levine Cancer Institute Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve SC, Cleveland, Ohio
  - Northwest Cancer Specialists Portland Loc, Portland, Oregon
  - St. Luke's Hospital and Health Network St Luke's (2), Bethlehem, Pennsylvania
  - Charleston Hematology Oncology Association PA, Charleston, South Carolina
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Vanderbilt University Medical Center Vanderbilt - Thompson Ln, Nashville, Tennessee
  - Texas Oncology P A Midtown, Dallas, Texas
  - Texas Oncology P A TX Onc - Bedford, Dallas, Texas
  - Texas Oncology P A TX Onc - Med City Dallas, Dallas, Texas
  - Texas Oncology P A TX Onc - Southwest, Dallas, Texas
  - Oncology Consultants Oncology Consultants, P.A., Houston, Texas
  - Cancer Therapy and Research Center UT Health Science Center Institute for Drug Development, San Antonio, Texas
  - Utah Cancer Specialists Dept.of Utah Cancer Spec. (3), Salt Lake City, Utah
  - Oncology Hematology Associates of Southeast Virginia Salem VA Branch, Roanoke, Virginia
  - Kadlec Clinic Hematology and Oncology Kadlec Clinic Hematology & Onc, Kennewick, Washington
  - West Virginia University/ Mary Babb Randolph Cancer Center Dept of Oncology, Morgantown, West Virginia
  - Cancer TEAM Bellin Health Belin Health, Green Bay, Wisconsin
  - Dean Health System Dean Hematology Oncology, Madison, Wisconsin
  - University of Wisconsin / Paul P. Carbone Comp Cancer Center Univ Wisc 3, Madison, Wisconsin
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Rio Negro, Viedma
- Australia (7):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Woollongong, New South Wales
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (3):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (7):
  - Novartis Investigative Site, Jette, Brussels Capital
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Wilrijk
- Brazil (7):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Ijuí, Rio Grande do Sul
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Sorocaba, São Paulo
- Canada (14):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Kelowna, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Laval, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Regina, Saskatchewan
- China (10):
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Shengyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Czechia (3):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Olomouc, CZE
  - Novartis Investigative Site, Brno
- France (18):
  - Novartis Investigative Site, Nice, Alpes Maritimes
  - Novartis Investigative Site, Dijon, Cote D Or
  - Novartis Investigative Site, Saint Priest En Jarez, Pays de la Loire Region
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (16):
  - Novartis Investigative Site, Langen, Hesse
  - Novartis Investigative Site, Recklinghausen, North Rhine-Westphalia
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Mühlhausen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Velbert
  - Novartis Investigative Site, Würzburg
- Greece (4):
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Szolnok
- Israel (5):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (17):
  - Novartis Investigative Site, Cuneo, CN
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Lido di Camaiore, LU
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Rimini, RN
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Mirano, VE
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Napoli
- Japan (12):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Sakyo Ku, Kyoto
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Koto Ku, Tokyo
- Novartis Investigative Site, Nijmegen, Netherlands
- Novartis Investigative Site, Surquillo, Lima region, Peru
- Poland (3):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Warsaw
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Košice
- South Africa (2):
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Parktown
- South Korea (3):
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Spain (16):
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Jaén, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Toledo, Castille-La Mancha
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, Las Palmas de Gran Canarias, Las Palmas de Gran Canaria
  - Novartis Investigative Site, San Sebastián de los Reyes, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Zaragoza
- Switzerland (3):
  - Novartis Investigative Site, Bellinzona
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Zurich
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Bangkok, Thailand
- United Kingdom (8):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Derby
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Campone M, Im SA, Iwata H, Clemons M, Ito Y, Awada A, Chia S, Jagiello-Gruszfeld A, Pistilli B, Tseng LM, Hurvitz S, Masuda N, Cortes J, De Laurentiis M, Arteaga CL, Jiang Z, Jonat W, Le Mouhaer S, Sankaran B, Bourdeau L, El-Hashimy M, Sellami D, Baselga J. Buparlisib plus fulvestrant versus placebo plus fulvestrant for postmenopausal, hormone receptor-positive, human epidermal growth factor receptor 2-negative, advanced breast cancer: Overall survival results from BELLE-2. Eur J Cancer. 2018 Nov;103:147-154. doi: 10.1016/j.ejca.2018.08.002. Epub 2018 Sep 18. PMID 30241001
- [Derived] Baselga J, Im SA, Iwata H, Cortes J, De Laurentiis M, Jiang Z, Arteaga CL, Jonat W, Clemons M, Ito Y, Awada A, Chia S, Jagiello-Gruszfeld A, Pistilli B, Tseng LM, Hurvitz S, Masuda N, Takahashi M, Vuylsteke P, Hachemi S, Dharan B, Di Tomaso E, Urban P, Massacesi C, Campone M. Buparlisib plus fulvestrant versus placebo plus fulvestrant in postmenopausal, hormone receptor-positive, HER2-negative, advanced breast cancer (BELLE-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2017 Jul;18(7):904-916. doi: 10.1016/S1470-2045(17)30376-5. Epub 2017 May 30. PMID 28576675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 274 centers in 29 countries worldwide (Argentina, Australia, Austria, Belgium, Brazil, Canada, China, Czech Republic, France, Germany, Greece, Hungary, Israel, Italy, Japan, Republic of Korea, The Netherlands, Peru, Poland, Russia, Singapore, Slovakia, South Africa, Spain, Switzerland, Taiwan, Thailand, UK and USA.).
Pre-assignment Details: Approximately 1200 patients were planned to be enrolled in the study. A total of 1147 patients were randomized and analyzed (576 in the buparlisib + fulvestrant and 571 in the placebo + fulvestrant arm). Not completed: in Randomization Phase=Randomized and not Treated; in Treatment Phase=Discontinued study treatment per Protocol.
Period: Randomization Phase
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Started (All randomized patients (FAS)) | 576 | 571
Safety Set (SS) (At least 1 dose of study treatment and a 1 post baseline safety assessment) | 573 | 570
Completed (Randomized and treated) | 574 | 569
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Death | 0 | 1
Period: Treatment Phase
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Started (All patients in FAS that were treated) | 574 | 569
BKM120 Pharmacokinetic Analysis Set (At least one dose of Buparlisib and 1 evaluable buparlisib concentration measurement) | 93 | 0
Full Pharmacokinetic Analysis Set (FPAS) (A subset of the patients in the Buparlisib PAS) | 35 | 0
Completed | 0 | 0
Not Completed | 574 | 569
Not completed — Adverse Event | 80 | 12
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-compliance with Study Treatment | 8 | 1
Not completed — Physician Decision | 27 | 24
Not completed — Progressive Disease | 377 | 486
Not completed — Protocol Deviation | 2 | 3
Not completed — Study terminated by Sponsor | 18 | 15
Not completed — Subject/Guardian Decision | 55 | 23
Not completed — Death | 6 | 5
Period: Post-Treatment Efficacy Follow-Up Phase
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Started (All patients who discontinued treatment and entered Post-Treatment Efficacy Follow-Up Phase) | 89 (All patients who entered Post-Treatment Efficacy Fup Phase) | 29 (All patients who entered Post-Treatment Efficacy Fup Phase)
Completed | 0 | 0
Not Completed | 89 | 29
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 10 | 3
Not completed — Progressive Disease | 24 | 8
Not completed — Subject/Guardian Decision | 11 | 1
Not completed — Death | 4 | 4
Not completed — New therapy for study indication | 38 | 13

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant | Total
Number analyzed (Participants) | 576 | 571 | 1147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 329 | 378 | 707
  >=65 years | 247 | 193 | 440
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (10.20) | 60.6 (10.08) | 61.4 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 576 | 571 | 1147
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 132 | 153 | 285
  Black | 5 | 16 | 21
  Caucasian | 402 | 376 | 778
  Other | 18 | 7 | 25
  Unknown | 19 | 18 | 37
  Missing | 0 | 1 | 1
ECOG Performance Status [Count of Participants; unit: Participants]
  Grade 0 = No Restrictions | 333 | 344 | 677
  Grade 1 = Only Light Work | 231 | 211 | 442
  Grade 2 = Only Self Care | 11 | 16 | 27
  Grade 3 = Only Limited Self-Care | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on Local Investigator Assessment - Full Analysis Set (FAS) in Full Population, Main Study Cohort and PI3K Unknown Cohort
Description: Progression Free Survival (PFS) is defined as the time from date of randomization to the date of first radiologically documented progression or death due to any cause. If a patient did not progress or die at the time of the analysis data cut-off or start of new antineoplastic therapy, PFS was censored at the date of the last adequate tumor assessment before the earliest of the cut-off date or the start date of additional anti-neoplastic therapy. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria RECIST v1.1, as 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline and/or unequivocal progression of the non-target lesions and/or appearance of a new lesion. In addition to the relative increase of 20%, the sum must demonstrate an absolute increase of at least 5 mm.
Time Frame: Date of randomization to the date of first documented tumor progression or death from any cause, whichever occurs first, reported between day of first patient randomized up to approximately 4 years
Population: Full Analysis Set (FAS) in the Full Population, the Main Study Cohort (known PI3K pathway activation status [activated, non activated]) and the PI3K unknown cohort (PI3K pathway unknown status) were considered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 576 | 571
Months
  FAS-Full population | 6.9 [6.8 to 7.8] | 5.0 [4.0 to 5.2]
  FAS-Main cohort: number analyzed (Participants) | 427 | 424
  FAS-Main cohort | 6.8 [5.0 to 7.0] | 4.5 [3.3 to 5.0]
  FAS-PI3K pathway activated: number analyzed (Participants) | 188 | 184
  FAS-PI3K pathway activated | 6.8 [4.9 to 7.1] | 4.0 [3.1 to 5.2]
  FAS-PI3K pathway non-activated: number analyzed (Participants) | 239 | 240
  FAS-PI3K pathway non-activated | 6.9 [4.6 to 7.2] | 4.6 [3.3 to 5.1]
  FAS-PI3K pathway unknown: number analyzed (Participants) | 149 | 147
  FAS-PI3K pathway unknown | 8.7 [7.0 to 12.4] | 6.8 [5.0 to 8.4]
Statistical Analysis 1: Comparison: BKM120 100mg + Fulvestrant vs Placebo + Fulvestrant; FAS-Full population; Test type: Other — Comparison of progression-free survival (PFS) (based on local investigator assessment) between the two treatment groups using a stratified log-rank test at one-sided 2.5% level of significance; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.67 to 0.89]
Statistical Analysis 2: Comparison: BKM120 100mg + Fulvestrant vs Placebo + Fulvestrant; FAS-Main cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.003, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.68 to 0.94]
Statistical Analysis 3: Comparison: BKM120 100mg + Fulvestrant vs Placebo + Fulvestrant; FAS-PI3K pathway activated; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.015, Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.60 to 0.97]
Statistical Analysis 4: Comparison: BKM120 100mg + Fulvestrant vs Placebo + Fulvestrant; FAS-PI3K pathway non-activated; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.67 to 1.03]
Statistical Analysis 5: Comparison: BKM120 100mg + Fulvestrant vs Placebo + Fulvestrant; FAS-PI3K pathway unknown; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.52 to 0.94]

2. Secondary Outcome: Overall Survival (OS) - Full Analysis Set (FAS) in Full Population, Main Study Cohort and PI3K Unknown Cohort
Description: Overall Survival (OS) is defined as the time from date of randomization to date of death due to any cause. If a patient was not known to have died by the date of analysis cut-off, OS was censored at the date of last known date patient alive. Patients were followed up for the duration of the study and for an expected average of every 3 months after end of treatment.
Time Frame: Every 3 months following end of treatment visit, assessed for approximately 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 576 | 571
Months
  FAS-Full population | 33.2 [30.0 to 37.3] | 30.4 [27.9 to 32.2]
  FAS-Main cohort: number analyzed (Participants) | 427 | 424
  FAS-Main cohort | 30.9 [25.1 to 35.4] | 28.9 [25.9 to 31.1]
  FAS-PI3K pathway activated: number analyzed (Participants) | 188 | 184
  FAS-PI3K pathway activated | 33.6 [23.8 to 40.0] | 27.5 [24.4 to 31.3]
  FAS-PI3K pathway non-activated: number analyzed (Participants) | 239 | 240
  FAS-PI3K pathway non-activated | 28.8 [23.0 to 33.2] | 30.0 [26.0 to 33.4]
  FAS-PI3K pathway unknown: number analyzed (Participants) | 149 | 147
  FAS-PI3K pathway unknown | 42.3 [36.5 to NA] — NA: Not estimable due to insufficient number of participants with events | 36.0 [31.0 to 43.5]
Statistical Analysis 1: Comparison: BKM120 100mg + Fulvestrant vs Placebo + Fulvestrant; FAS-Full population; Test type: Other — Comparison of overall survival (OS) (based on local investigator assessment) between the two treatment groups using a stratified log-rank test at one-sided 2.5% level of significance; p = 0.045, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.74 to 1.02]
Statistical Analysis 2: Comparison: BKM120 100mg + Fulvestrant vs Placebo + Fulvestrant; FAS-Main cohort; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.144, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.75 to 1.09]
Statistical Analysis 3: Comparison: BKM120 100mg + Fulvestrant vs Placebo + Fulvestrant; FAS-PI3K pathway activated; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.61 to 1.08]
Statistical Analysis 4: Comparison: BKM120 100mg + Fulvestrant vs Placebo + Fulvestrant; FAS-PI3K pathway non-activated; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.77 to 1.24]
Statistical Analysis 5: Comparison: BKM120 100mg + Fulvestrant vs Placebo + Fulvestrant; FAS-PI3K pathway unknown; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.52 to 1.06]

3. Secondary Outcome: Overall Response Rate (ORR) - Full Analysis Set (FAS) in Full Population, Main Study Cohort and PI3K Unknown Cohort
Description: Overall Response Rate (ORR) is defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR) based on local investigator's assessment according to RECIST 1.1. ORR was analyzed in the full population. Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for target/non target lesions: Complete Response (CR), disappearance of all target/non target lesions (all lymph nodes assigned as non-target lesions must be non-pathological in size (< 10 mm short axis)); Partial response (PR), >=30% decrease in the sum of the longest diameter of target lesions ; Overall Response (OR)= CR+PR. Only descriptive analysis performed.
Time Frame: From the date of randomization until the date of the first documented disease progression or date of death from any cause whichever came first, assessed for approximately 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 576 | 571
Percentage of Participants
  FAS-Full population | 11.8 [9.3 to 14.7] | 7.7 [5.7 to 10.2]
  FAS-Main cohort: number analyzed (Participants) | 427 | 424
  FAS-Main cohort | 11.0 [8.2 to 14.4] | 7.8 [5.4 to 10.8]
  FAS-PI3K pathway activated: number analyzed (Participants) | 188 | 184
  FAS-PI3K pathway activated | 10.6 [6.6 to 16.0] | 8.2 [4.6 to 13.1]
  FAS-PI3K pathway non-activated: number analyzed (Participants) | 239 | 240
  FAS-PI3K pathway non-activated | 11.3 [7.6 to 16.0] | 7.5 [4.5 to 11.6]
  FAS-PI3K pathway unknown: number analyzed (Participants) | 149 | 147
  FAS-PI3K pathway unknown | 14.1 [8.9 to 20.7] | 7.5 [3.8 to 13.0]

4. Secondary Outcome: Clinical Benefit Rate (CBR) - Full Analysis Set (FAS) in Full Population, Main Study Cohort and PI3K Unknown Cohort
Description: Clinical Benefit Rate (CBR) is defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) or stable disease (SD) or Non-CR/non-PD lasting more than 24 weeks based on local investigator's assessment according to RECIST 1.1. CBR was analyzed in the full population. Only descriptive analysis performed.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 576 | 571
Percentage of Participants
  FAS-Full population | 43.8 [39.7 to 47.9] | 42.0 [37.9 to 46.2]
  FAS-Main cohort: number analyzed (Participants) | 427 | 424
  FAS-Main cohort | 41.7 [37.0 to 46.5] | 39.6 [34.9 to 44.5]
  FAS-PI3K pathway activated: number analyzed (Participants) | 188 | 184
  FAS-PI3K pathway activated | 40.4 [33.3 to 47.8] | 40.8 [33.6 to 48.2]
  FAS-PI3K pathway non-activated: number analyzed (Participants) | 239 | 240
  FAS-PI3K pathway non-activated | 42.7 [36.3 to 49.2] | 38.8 [32.6 to 45.2]
  FAS-PI3K pathway unknown: number analyzed (Participants) | 149 | 147
  FAS-PI3K pathway unknown | 49.7 [41.4 to 58.0] | 49.0 [40.7 to 57.3]

5. Secondary Outcome: Number of Participants With On-Treatments Adverse Events, Serious Adverse Events and Deaths
Description: Analysis of frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths. Only descriptive analysis performed.
Time Frame: From first dose of study treatment to 30 days after last dose of study treatment, assessed for approximately 5 years
Population: Safety Set (SS) in Full Population
Measure: Count of Participants; unit: Participants
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 573 | 570
Participants
  On-treatment Adverse Event (AEs) | 569 | 532
  On-treatment Serious Adverse Event (SAEs) | 144 | 101
  On-treatment Deaths | 12 | 13
  Primary cause of Death = Study Indication | 6 | 7
  Primary cause of Death = Unknown reason | 2 | 0
  Primary cause of Death = Disease Progression | 2 | 2
  Primary cause of Death = Pneumonia | 1 | 0
  Primary cause of Death = Septic Shock | 1 | 0
  Primary cause of Death = Cerebral Haemorrhage | 0 | 1
  Primary cause of Death = Cerebral Accident | 0 | 1
  Primary cause of Death = Sudden Death | 0 | 1
  Primary cause of Death = Urosepsis | 0 | 1

6. Secondary Outcome: Plasma Concentration-time Profiles of BKM120 in Combination With Fulvestrant at Cycle 2 Day 1
Description: Plasma samples were collected from the first 200 BKM120-treated patients on Cycle 2 Day 1 (at pre-dose, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h and 24h [before Cycle 2 Day 2 dose] post-dose). Each cycle is 28 days. Only descriptive analysis performed.
Time Frame: Cycle2 Day1 (0, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours post-dose). Each cycle is 28 days.
Population: Full Pharmacokinetic Analysis Set (FPAS) included the subset of the patients in the buparlisib PAS who:
  * Received all planned doses of BKM120 100mg + Fulvestrant preceding full PK profile assessment
  * Did not vomit within 4 hours of buparlisib dosing after administration
  * Had an evaluable full PK profile available
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | BKM120 100mg + Fulvestrant
Number analyzed (Participants) | 35
nanogram per milliliter (ng/mL)
  C2D1 0hr (predose) | 768.306 (69.1)
  C2D1 0.5hr: number analyzed (Participants) | 34
  C2D1 0.5hr | 750.767 (55.4)
  C2D1 1hr | 988.341 (49.2)
  C2D1 1.5hr | 1082.086 (45.0)
  C2D1 2hr | 1099.517 (36.4)
  C2D1 3hr: number analyzed (Participants) | 34
  C2D1 3hr | 1081.123 (43.2)
  C2D1 4hr | 935.485 (43.0)
  C2D1 6hr | 795.555 (45.1)
  C2D1 8hr: number analyzed (Participants) | 34
  C2D1 8hr | 808.886 (50.5)
  C2D1 24hr: number analyzed (Participants) | 34
  C2D1 24hr | 712.336 (52.7)

7. Secondary Outcome: Predose Trough Concentration-time Profile of BKM120 in Combination With Fulvestrant Over Time - Pharmacokinetic Analysis Set (PAS)
Description: Pre-dose samples were collected for trough concentrations at Cycle 2 Day 1, Cycle 2 Day 15 and Cycle 3 Day 1. Each cycle is 28 days. Only descriptive analysis performed.
Time Frame: Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1. Each cycle is 28 days.
Population: BKM120 Pharmacokinetic Analysis Set or Buparlisib pharmacokinetic analysis set (Buparlisib PAS) included all patients who received at least one dose of study medication buparlisib and had at least one evaluable post-treatment buparlisib concentration measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | BKM120 100mg + Fulvestrant
Number analyzed (Participants) | 93
nanogram per milliliter (ng/mL)
  Cycle 2 Day 1: number analyzed (Participants) | 69
  Cycle 2 Day 1 | 733.278 (75.6)
  Cycle 2 Day 15: number analyzed (Participants) | 23
  Cycle 2 Day 15 | 735.172 (51.2)
  Cycle 3 Day 1: number analyzed (Participants) | 31
  Cycle 3 Day 1 | 716.414 (84.8)

8. Secondary Outcome: Median Time to Definitive Deterioration of the ECOG Performance Status - Full Analysis Set (FAS)
Description: Time to definitive deterioration of the ECOG PS was defined as the time between the date of randomization and the date of the assessment at which definitive deterioration was seen. Only descriptive analysis performed.
Time Frame: Up to approx 27 months
Population: Full Analysis (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 576 | 571
Months | 24.0 [17.1 to NA] — NA: Not Estimable due to number of events censored | 26.4 [19.9 to NA] — NA: Not Estimable due to number of events censored

9. Secondary Outcome: Health-related Quality of Life (HRQoL):Time to 10% Definitive Deterioration in the Global Health Status/Quality of Life Per EORTC-QLQ-C30
Description: The global health status/QoL scale score of the QLQ-C30 is identified as the primary PRO variable of interest. Physical Functioning (PF), Emotional Functioning (EF) and Social Functioning (SF) scale scores of the QLQ-C30. The time to definitive 10% deterioration is defined as the time from the randomization date to the date of an event, which is defined as a worsening (decrease) in score by at least 10% compared to baseline, with no later increase above this threshold observed during the course of the study or death due to any cause. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high /healthy level of functioning, a high score for the global health status / QoL represents a high QoL. Patients were assessed up to approx. 8.3 months. Only descriptive analysis performed.
Time Frame: Cycle 1 day 1, cycle 1 day 15, 6 weeks after randomisation and then every 8 weeks until end of treatment
Population: Full Analysis (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 576 | 571
Months | 7.10 [6.01 to 9.82] | 11.50 [8.80 to 14.32]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, assessed for approximately 5 years
Description: Any sign or symptom that occurs during the study treatment and 30 days post treatment follow up.
  Maximum exposure to study treatments = 52.9 months (BKM120 100mg + Fulvestrant treatment group) and 69.6 months (Placebo + Fulvestrant treatment group).
Groups:
- BKM120 100 mg + Fulvestrant: BKM120 100 mg per day and fulvestrant given until progression or as described in the protocol.
Arm/Group | BKM120 100 mg + Fulvestrant | Placebo + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 12/573 | 13/570
Serious Adverse Events (participants affected / at risk) | 146/573 | 101/570
Other Adverse Events (participants affected / at risk) | 560/573 | 485/570
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 100 mg + Fulvestrant (N=573) | Placebo + Fulvestrant (N=570)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 2
Cataract (Eye disorders) | 1 | 0
Retinal tear (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 2
Obstruction gastric (Gastrointestinal disorders) | 2 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Stomatitis (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 5
Asthenia (General disorders) | 7 | 2
Breakthrough pain (General disorders) | 1 | 0
Condition aggravated (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 7 | 0
General physical health deterioration (General disorders) | 6 | 2
Incarcerated hernia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Sudden death (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Candida sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Infectious colitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 2 | 2
Peritonitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 3 | 5
Pyelonephritis (Infections and infestations) | 0 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyuria (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 1 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 1
Urosepsis (Infections and infestations) | 1 | 2
Vestibular neuronitis (Infections and infestations) | 0 | 1
Viral labyrinthitis (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 3 | 3
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 17 | 1
Aspartate aminotransferase increased (Investigations) | 14 | 1
Blood bilirubin increased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 2 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Coordination abnormal (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 3
Dizziness (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Movement disorder (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 2
Status epilepticus (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 4
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 2 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Vascular dementia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 4 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 100 mg + Fulvestrant (N=573) | Placebo + Fulvestrant (N=570)
Anaemia (Blood and lymphatic system disorders) | 38 | 51
Abdominal pain (Gastrointestinal disorders) | 40 | 30
Abdominal pain upper (Gastrointestinal disorders) | 46 | 38
Constipation (Gastrointestinal disorders) | 68 | 71
Diarrhoea (Gastrointestinal disorders) | 198 | 84
Dry mouth (Gastrointestinal disorders) | 46 | 20
Dyspepsia (Gastrointestinal disorders) | 52 | 25
Nausea (Gastrointestinal disorders) | 227 | 138
Stomatitis (Gastrointestinal disorders) | 124 | 40
Vomiting (Gastrointestinal disorders) | 92 | 79
Asthenia (General disorders) | 113 | 62
Fatigue (General disorders) | 187 | 143
Injection site pain (General disorders) | 27 | 34
Oedema peripheral (General disorders) | 38 | 30
Pyrexia (General disorders) | 44 | 22
Upper respiratory tract infection (Infections and infestations) | 29 | 31
Urinary tract infection (Infections and infestations) | 46 | 31
Alanine aminotransferase increased (Investigations) | 229 | 39
Aspartate aminotransferase increased (Investigations) | 217 | 55
Blood alkaline phosphatase increased (Investigations) | 40 | 31
Gamma-glutamyltransferase increased (Investigations) | 45 | 39
Weight decreased (Investigations) | 84 | 24
Decreased appetite (Metabolism and nutrition disorders) | 174 | 68
Hyperglycaemia (Metabolism and nutrition disorders) | 244 | 46
Hypokalaemia (Metabolism and nutrition disorders) | 41 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 62 | 74
Back pain (Musculoskeletal and connective tissue disorders) | 66 | 72
Bone pain (Musculoskeletal and connective tissue disorders) | 38 | 34
Muscle spasms (Musculoskeletal and connective tissue disorders) | 32 | 21
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 27 | 40
Pain in extremity (Musculoskeletal and connective tissue disorders) | 51 | 61
Dizziness (Nervous system disorders) | 75 | 30
Dysgeusia (Nervous system disorders) | 84 | 22
Headache (Nervous system disorders) | 88 | 79
Tremor (Nervous system disorders) | 44 | 7
Anxiety (Psychiatric disorders) | 129 | 53
Depression (Psychiatric disorders) | 152 | 56
Insomnia (Psychiatric disorders) | 60 | 50
Mood altered (Psychiatric disorders) | 40 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 76 | 69
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 | 56
Alopecia (Skin and subcutaneous tissue disorders) | 41 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 69 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 88 | 33
Rash (Skin and subcutaneous tissue disorders) | 187 | 39
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 39 | 8
Hot flush (Vascular disorders) | 33 | 53
Hypertension (Vascular disorders) | 57 | 29

LIMITATIONS AND CAVEATS:
Novartis made the decision not to pursue further development of buparlisib and to terminate the ongoing studies in Breast Cancer. The CBKM120F2302 study was terminated on 19-Apr-2019 (last subject last visit).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.